CLINICAL TRIAL: NCT01426035
Title: Phase III of Safety and Efficacy Study of Topic Mucopolysaccharide Polysulfate Cream 5mg/g in the Superficial Varicose Veins Treatment
Brief Title: Safety And Efficacy Study Of Topic Mucopolysaccharide Polysulfate Cream In The Superficial Varicose Veins Treatment
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MPSEMS0110_cream
Record Dates: First submitted 2011-05-09; First posted 2011-08-30 (Estimated); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: VARICOSE VEINS
Keywords: SUPERFICIAL VARICOSE VEINS
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GROUP 1 (Experimental)
  Interventions: Drug: TOPIC MUCOPOLYSACCHARIDE POLYSULFATE CREAM 5MG/G
- GROUP 2 (Active Comparator)
  Interventions: Drug: TOPIC MUCOPOLYSACCHARIDE POLYSULFATE CREAM 5MG/G

INTERVENTIONS:
Drug: TOPIC MUCOPOLYSACCHARIDE POLYSULFATE CREAM 5MG/G — APLIED 4 TIMES/DAY AT LESION

SUMMARY:
Evaluate the safety, tolerability and effectiveness of mucopolysaccharide polysulfate cream in the treatment of superficial varicose veins

ELIGIBILITY:
Inclusion Criteria:

* Patients must be able to understand the study procedures, agree to participate, and give written consent.
* Patients must be able to follow the study medication regimen.
* Patients with inflammatory process in superficial veins for more than 72 hours.
* Presence of symmetric lesions to compare one side to the other.

Exclusion Criteria:

* Pregnancy or risk of pregnancy.
* Lactation.
* Use of topical or systemic anti-inflammatory, antihistamine or immunosuppressive drugs within the last 48 hours prior to the study
* Any alteration at other deep veins.
* History of atopy or allergic diseases.
* History of allergy to any component of the formulations.
* Other conditions considered by the investigator as reasonable for non-eligibility

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2014-12 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Efficacy - Symptoms reduction | Evaluation time: 15 days treatment
  The primary outcome measure will be evaluated for: Lesion area reduction, reduction of symptoms time and edema

SECONDARY OUTCOMES:
Efficacy - patient evaluation | Evaluation time: 15 days treatment
  The secondary outcome measure will be measured by subjective opinion (daily register).

CONTACTS AND LOCATIONS:
Overall Officials: FLAVIA ADDOR, Principal Investigator — Medcin Instituto da Pele; Felipe Pinho, MD, Study Director — EMS
Locations (1):
- Medcin Instituto Da Pele, Osasco, São Paulo, Brazil